CLINICAL TRIAL: NCT02777242
Title: An Open-Label Study to Evaluate the Safety of Testosterone Enanthate After Two Single-Dose Injections Via QuickShot® Testosterone by Intended Users and QuickShot™ Summative Usability Study
Brief Title: Safety of Subcutaneous Testosterone Enanthate in Adult Male Hypogonadism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Antares Pharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QST-16-006
Record Dates: First submitted 2016-05-12; First posted 2016-05-19 (Estimated); Results first posted 2018-02-26 (Actual); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: Hypogonadism
Keywords: Hypogonadism; Testosterone enanthate
MeSH Terms: conditions — Hypogonadism | interventions — Testosterone; testosterone enanthate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Testosterone enanthate auto-injector (Experimental): Testosterone enanthate administered subcutaneously once each week. Auto-injection of QST 50 mg or 75 mg or 100 mg [Device: QuickShot® Testosterone (QST)]
  Interventions: Combination Product: Testosterone enanthate auto-injector

INTERVENTIONS:
Combination Product: Testosterone enanthate auto-injector — SC injections of QST 50 mg or 75 mg or 100 mg
  Other Names: Testosterone; Testosterone enanthate; QuickShot® Testosterone (QST)

SUMMARY:
Evaluation of the safety and tolerability of testosterone enanthate (TE) following a single dose via QuickShot® Testosterone (QST) when administered by intended users in a usability study.

DETAILED DESCRIPTION:
Intended users are patients as well as patient caregivers, such as family members or friends who are able to assist the patient to administer the medication (i.e. lay users). One user group of approximately 15 patients will have their dose administered by a qualified healthcare professional (HCP).

ELIGIBILITY:
Inclusion Criteria

Each patient must meet all of the following criteria at screening to participate in the study:

1. The patient is 18 years of age or older;
2. The patient speaks, reads, and understands the English language at a sixth grade reading level or higher;
3. The patient is willing to have photographs taken and/or be video recorded while he completes study tasks, which will be de-identified prior to any potential use of the image(s) for scientific or educational purposes;
4. The patient has sufficient availability to participate in the study and to comply with the study schedule;
5. The patient has his own transportation to and from the study site;
6. The patient demonstrates the ability to understand and the willingness to follow all study instructions; and
7. The patient has read, stated he understands, and has signed the Informed Consent Form (ICF).
8. The patient has been diagnosed with hypogonadism;
9. The patient is a male;
10. The patient has a documented history of hypogonadism. Diagnosis must include documentation of consistent signs and symptoms of androgen deficiency;
11. Patients in good health as determined by the Investigator and based on medical history, physical examination, vital signs, electrocardiogram (ECG), and clinical laboratory tests;
12. All male patients must practice effective contraception during the study and for 30 days after receiving the last dose of study drug. Acceptable methods of birth control include condom with spermicide, vasectomy, or monogamous relations with a female partner who is of non child-bearing potential (post-menopausal, surgical, or congenital sterility) or is of child bearing potential and practicing a reliable method of contraception (hormonal contraception, double barrier methods with spermicide, or intrauterine device); and
13. Patients must have the ability to provide written informed consent and comply with all study requirements and restrictions including the study visit schedule.

Exclusion Criteria

Patients will be excluded from participation in the study if any of the following criteria apply:

1. Failure to meet 1 or more Inclusion Criterion;
2. The patient has participated in interviews, focus groups, or studies for any medical products or therapies within the past 3 months or in a prior QST auto-injector usability study, clinical trial, and/or has previous exposure to the investigational device;
3. The patient or someone he lives with works or has worked for a Marketing/Market Research Company, pharmaceutical or medical device company, a manufacturer, distributor, or wholesaler of non-prescription drug products, or a government health agency;
4. Individuals who have had an allergic reaction or idiosyncratic reaction to sesame seeds, sesame products, and/or sesame oil;
5. History of food anaphylaxis;
6. History of intolerance, allergy, or idiosyncratic reaction to testosterone products;
7. Unstable psychiatric illnesses;
8. Lifetime history of psychosis, suicidal behavior, bipolar disorder, or personality disorder; active suicidal ideation within 6 months prior to screening; or inadequately treated depression. Note: Patients with depression who have been adequately treated and with stable response for 3 months may be admitted into the study at the Investigator's discretion;
9. Body mass index 40 kg/m2;
10. Hematocrit 52% at Initial Screening Visit;
11. Individual history or current evidence of breast or prostate cancer;
12. Other malignancy diagnosed or treated within 5 years of the date of Initial Screening Visit with the exception of non-melanoma carcinoma of the skin;
13. Elevated prostate-specific antigen (PSA) for age. Prostate-specific antigen 2.5 ng/mL in men 18 to 60 years old and 4 ng/mL in men 61 years and older is exclusionary;
14. Presence of prostate nodule or induration upon digital rectal exam;
15. Obstructive uropathy of prostatic origin and of a severity that, in the opinion of the Investigator, contraindicates the use of testosterone;
16. Patients with poorly controlled diabetes. Patients on a stable dose and regimen of anti diabetic medications for a minimum of 4 weeks, and who have a hemoglobin A1c level of 7.5% may participate in the study;
17. Patients with New York Heart Association Class III or IV congestive heart failure;
18. Within 6 months of the Initial Screening Visit, have had myocardial infarction, unstable angina leading to hospitalization, percutaneous coronary intervention, coronary artery bypass graft, uncontrolled cardiac arrhythmia, stroke transient ischemia attack, carotid revascularization, endovascular procedure, or surgical intervention for peripheral vascular disease;
19. History of, or current treatment for, thromboembolic disease or current use of anti thromboembolic medications. Use of low-dose aspirin is permitted for routine cardioprophylaxis;
20. Patients intermittently taking adrenocorticotropic hormone, oral, or depot corticosteroids (ongoing regimens required for panhypopituitarism or adrenal failure are permitted);
21. Untreated sleep apnea;
22. Historical or current evidence of any clinically significant disease or disorder that, in the judgment of the Investigator, may cause participation in this study to be detrimental to the patient or which may influence the results of the study. This includes cardiovascular, renal, hepatic, hematological, endocrine, gastrointestinal, or pulmonary disease;
23. Positive serology for human immunodeficiency virus antibodies, hepatitis B surface antigen, or hepatitis C virus antibody at the Initial Screening Visit;
24. Current evidence of alcohol or drug abuse. A positive drug screen is exclusionary without documentation of a current prescription and medical condition requiring treatment with the drug for which the screen is positive. Exception: tetrahydrocannabinol is allowed in states where recreational use of marijuana is legal;
25. Any skin condition that could confound injection site assessments (eg, dermatographism, urticaria, or atopic dermatitis). Tattoos, scarring, or psoriasis of the injection site is prohibited;
26. Administration of any other investigational compound within 1 month prior to Initial Screening Visit or 5 half-lives of the investigational product (whichever is longer);
27. Patients considering or scheduled to undergo any major surgery or dental procedure anticipated to be associated with significant blood loss (500 mL) during the study;
28. Systolic blood pressure (SBP) 140 mmHg and/or diastolic blood pressure (DBP) 90 mmHg at the Initial Screening Visit. Patients with treated hypertension and SBP 140 and/or DBP 90 mmHg at the Initial Screening Visit must be on a stable dose of antihypertensive medication for at least 14 days at Day -1 (Baseline Visit) and plan to remain on the same dose throughout the duration of the study; or
29. Unable to understand verbal or written English or any other language in which a certified translation of the informed consent is available.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jed Kaminetsky, MD, Principal Investigator — Manhattan Medical Research
Locations (3):
- United States (3):
  - Birmingham, Alabama
  - New York, New York
  - Columbus, Ohio

RESULTS

PARTICIPANT FLOW:
Recruitment Details: In total, 66 patients were enrolled, of which 65 patients were randomized and were included in the Safety Population.
Pre-assignment Details: The Safety Population included all patients who were randomized and took at least one dose of Investigational Product. The Safety Population was used as the denominator in percentage calculations.
Groups:
- Testosterone Enanthate Auto-injector: Testosterone enanthate administered subcutaneously once each week via auto-injector of QST 50 mg or 75 mg or 100 mg [Device: QuickShot® Testosterone (QST)]
Period: Overall Study
Arm/Group | Testosterone Enanthate Auto-injector
Started | 65
Completed | 59
Not Completed | 6
Not completed — Other | 2
Not completed — Lost to Follow-up | 1
Not completed — Multiple | 1
Not completed — Sponsor's request | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Testosterone Enanthate Auto-injector
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.3 (8.98)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 65
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 17
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Adverse Events Receiving Testosterone Enanthate Via QST Auto-injector.
Description: Intended users were patients experiencing an adverse event that was considered to be a TEAE if the adverse event started on or after randomization, or existed prior to randomization and worsened in severity or relatedness to QST (QuickShot® Testosterone auto-injector) after randomization.
Time Frame: 3 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Testosterone Enanthate Auto-injector
Number analyzed (Participants) | 65
Participants
  Patients with any TEAE | 5
  Patients with any TEAE related to QST | 1
  Patients with SAE | 0
  Patients with TEAE leading to discontinuation | 0
  Patients with QST related TEAE and discontinuation | 0

ADVERSE EVENTS:
Time Frame: 3 Weeks
Description: An adverse event was considered to be a TEAE if the adverse event started on or after randomization, or existed prior to randomization and worsened in severity or relatedness to IP after randomization
Arm/Group | Testosterone Enanthate Auto-injector
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 5/65
OTHER ADVERSE EVENTS (reported when occurring in more than 1.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Testosterone Enanthate Auto-injector (N=65)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1)
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other